CLINICAL TRIAL: NCT06275321
Title: Physical Exercise Benefits in Breast Cancer Patients Undergoing Treatment
Brief Title: Physical Exercise Benefits for Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Principal Investigator, Elena Garcia Roca, Principal investigator, Universitat Jaume I
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Elena Garcia Roca
Record Dates: First submitted 2024-01-30; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Cancer, Breast; Sports Physical Therapy
Keywords: Oncology; Quality of live; Physical exercise; Physical activity; Physical fitness
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: A prospective ramonized clinical trial with two groups
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous-supervised online home-baased group (Experimental): Group following a supervised exercise program with an exercise cancer specialist
  Interventions: Other: Synchronous-supervised online home-based group
- Exercise recommendation group (Active Comparator): Group following general recommendations of physical exercise
  Interventions: Other: Exercise recommendation group

INTERVENTIONS:
Other: Synchronous-supervised online home-based group — An online exercise program combining endurance and strength training
  Arms: Synchronous-supervised online home-baased group
Other: Exercise recommendation group — General recommendation about physical exercise. No supervised
  Arms: Exercise recommendation group

SUMMARY:
The purpose of the study was to analyze the effect of a synchronous-supervised online home-based group during a 6-month exercise program on physical fitness, body composition and adherence compared to an exercise recommendation group of patients undergoing breast cancer treatment without supervision.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Diagnosted with breast cancer
* Undergoing cancer treatment
* No medical contraindications

Exclusion Criteria:

* Medical contraindications for sport practice
* Refusal to participate in the study
* Comorbilities

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer females undergoing cancer treatment
Enrollment: 60 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-07-27 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Cardiorrespiratory fitness | 24 weeks
  6 minutes walking test was performed in a 50 meter circuit. Meters completed during 6 minutes were recorded.
Strength - Chair Stand (repetitions) | 24 weeks
  Chair stand test was performed. Number of repetitions performed during 30 seconds was recorded.
Flexibility | 24 weeks
  Sit and Reach (centimeters): sitted and with stretched legs, the patient has to move a piece of wood on a bench. The centimeters moved by the patients are recorded
Incidence of treatments on quality of live assessed by EORTIC QLQ-C30 | 24 weeks
  QLQ-C30 questionnaire with 30 items was used to record the quality of life of the patients. Each item has a scale from 1 to 4, being 1 the lowest and 4 the highest outcome.
Adherence | 24 weeks
  Minutes on each training session were recorded to control the adherence.
Rating of perceived exertion | 24 weeks
  A Borg Scale (1-10) was used to control the intensity of the sessions, being 1 the lowest intensity and 10 the highest intensity.
Strength - Hand Grip (Kilograms) | 24 weeks
  Hand Grip (kilograms): a dynamometer (Grip Strength Dynamometer, Takker TKK, Tokio, Japón) was used to record hand grip.
Strength - Squat Jump (height in centimeters) | 24 weeks
  Squat Jump (centimeters): a contact platform (Chronojump Boscosystem, Barcelona, Spain) was used to record the height of the jump in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: M. Elena Garcia-Roca, MSc, Principal Investigator — Universitat Jaume I; Eladio J. Collado-Boira, PhD, Study Director — Universitat Jaume I
Locations (1):
- Jaume I University, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No